CLINICAL TRIAL: NCT06572137
Title: Prevalence of Parental Burnout Among Mothers of Children With Cerebral Palsy: Cross Sectional Study
Brief Title: Prevalence of Parental Burnout Among Mothers of Children With Cerebral Palsy
Status: Recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud khattab Ahmed eltohami Khalil, principal investigator, Cairo University
Other Study IDs: Mahmoud-005248
Record Dates: First submitted 2024-08-23; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Parents; Burnout; Children, Only; Cerebral Palsy
MeSH Terms: conditions — Burnout, Psychological; Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will be done to determine the prevalence of Parental Burnout among mothers of children with cerebral palsy.

Determine the relation between Parental Burnout syndrome and the motor function levels of children with cerebral palsy.

DETAILED DESCRIPTION:
Cerebral palsy is a significant physical disability in children, affecting 2-5 children per 1,000 live births globally. The prevalence varies between countries and is higher in low- and middle-income countries. Studies suggest a relationship between children's motor impairment and parental stress, which can lead to illness, negative family dynamics, and neglect. Parenting stress and pressure have increased, leading to exhaustion and burnout among parents. This study aims to investigate the prevalence of Parental Bowel Syndrome among mothers of children with CP and its relation to motor function levels.

ELIGIBILITY:
Inclusion Criteria:

* Mothers of children with CP of any age.
* Children diagnosed with CP.
* The age of children will range from 3-18 years old.

Exclusion Criteria:

* Mothers who refuse to participate in the study.
* Mothers of more than one disabled child.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Mothers of children with cerebral palsy of any age.
Study Population: The estimated prevalence of burnout among mothers of children with cerebral palsy is 65% with expected prevalence 56%
Sampling Method: Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
assessment of 4 dimensions of burnout | at baseline
  The Lebanese translation of the Parental burnout questionnaire, a 23-item self-report, includes four subscales: Emotional Exhaustion, Contrast, Feelings of Being Fed Up, and Emotional Distancing. The questionnaire has Cronbach's alphas of.93,.93,.90, and.81 for the sub-scales and.96 for the global score.

SECONDARY OUTCOMES:
assessment of gross motor function | at baseline
  The Gross Motor Function Classification System (GMFCS) categorizes children into Level I, Level II, Level III, Level IV, and Level V. Level I children can walk, climb stairs, and perform gross motor skills, while Level II and III require assistance, while Level IV and V require manual wheelchair use.

CONTACTS AND LOCATIONS:
Locations (1):
- out-patient clinic, faculty of physical therapy, Cairo university, Giza, Egypt